CLINICAL TRIAL: NCT05823428
Title: Arthroscopic Biological Augmentation With Subacromial Bursa for Bursal Side Partial-thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist,Chief assistant, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Subacromial bursa Augmentation
Record Dates: First submitted 2023-03-21; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Partial Thickness Rotator Cuff Tears
Keywords: partial thickness; bursal side; rotator cuff; full thickness; subacromial bursa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotator cuff debridement + acromioplasty (Active Comparator): Group A was formed by performing rotator cuff debridement + acromioplasty in 18 patients.
  Interventions: Procedure: Rotator cuff debridement + acromioplasty
- Augmentation with subacromial bursa + acromioplasty (Active Comparator): Group B was formed by performing augmentation with subacromial bursa + acromioplasty in 22 patients.
  Interventions: Procedure: Augmentation with subacromial bursa + acromioplasty

INTERVENTIONS:
Procedure: Augmentation with subacromial bursa + acromioplasty — Two intervention was planned. Rotator cuff debridement + acromioplasty group is mentioned as Group A (18 patients) and augmentation with subacromial bursa + acromioplasty is Group B
  Arms: Augmentation with subacromial bursa + acromioplasty
Procedure: Rotator cuff debridement + acromioplasty — Two intervention was planned. Rotator cuff debridement + acromioplasty group is mentioned as Group A (18 patients) and augmentation with subacromial bursa + acromioplasty is Group B
  Arms: Rotator cuff debridement + acromioplasty

SUMMARY:
The investigators aimed to compare the results of acromioplasty + arthroscopic debridement and acromioplasty + augmentation with subacromial bursa.

ELIGIBILITY:
Inclusion Criteria:

* bursal side rotator cuff tears in MRI sections
* Patients whose pain does not go away despite NSAIDs and standardized physical therapy by the same physiotherapist applied for 3 months
* 25-50% or 3-6 mm rotator cuff tear (Ellman grade 2) on the bursal side

Exclusion Criteria:

* Previous surgery
* tears greater than 50% or 6 mm

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of biological augmentation with bursa using postoperative clinical scores and MRI. | 18 months
  Our Primary Outcome Measure is to investigate the effects of biological augmentation with subacromial bursa in arthroscopic bursal-sided partial thickness rotator cuff repair with postoperative MRI and functional scores with Constant-Murley and Ases scores.

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)